CLINICAL TRIAL: NCT00021294
Title: Phase IIB Randomized, Double-Blinded, Placebo Controlled Study to Evaluate the Safety and Efficacy of Topical Difluoromethylornithine (DFMO) With and Without a Topical Corticosteroid Cream (Triamcinolone 0.1%) in the Therapy of Actinic Keratoses (AK) on the Forearms
Brief Title: Eflornithine With or Without Triamcinolone in Preventing Nonmelanoma Skin Cancer in Patients With Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068767; P01CA027502 (NIH); UARIZ-HSC-0072; NCI-H01-0075
Record Dates: First submitted 2001-07-11; First posted 2004-02-16 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Non-melanomatous Skin Cancer; Precancerous/Nonmalignant Condition
Keywords: basal cell carcinoma of the skin; squamous cell carcinoma of the skin; actinic keratosis
MeSH Terms: conditions — Precancerous Conditions; Carcinoma, Basal Cell; Keratosis, Actinic | interventions — Eflornithine; Triamcinolone

INTERVENTIONS:
Drug: eflornithine
Drug: triamcinolone

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. Eflornithine with or without triamcinolone may be effective in preventing nonmelanoma skin cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of eflornithine with or without triamcinolone in preventing nonmelanoma skin cancer in patients who have actinic keratosis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the safety and efficacy of eflornithine (DFMO) vs placebo as chemoprevention of non-melanoma skin cancer in patients with moderate to heavy actinic keratosis (AK). II. Determine whether this drug reverses AK in these patients. III. Determine whether triamcinolone reduces DFMO-induced skin irritation in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are randomized to 1 of 4 treatment arms. Arm I: Patients receive eflornithine (DFMO) topically and triamcinolone topically to forearms once daily. Arm II: Patients receive DFMO and placebo topically as in arm I. Arm III: Patients receive placebo and triamcinolone topically as in arm I. Arm IV: Patients receive 2 placebos topically as in arm I. Treatment continues for 6 months in the absence of unacceptable toxicity. Patients are followed at 2 weeks.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of actinic keratosis At least 3 clinically visible lesions on each lower posterior forearm Lesions must be discrete and quantifiable No prior or concurrent skin cancer on forearms Prior skin cancer (other than melanoma) on an area other than the forearms allowed unless chronic recurrent lesions indicate immunosuppression Concurrent skin cancer on an area other than the forearms allowed if active lesion previously excised

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No serious concurrent illness No immunosuppression due to medication or disease No invasive cancer (including melanoma) within the past 5 years Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception at least 28 days prior to and during study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 5 years since prior systemic chemotherapy At least 6 months since prior fluorouracil (5-FU) to forearms Prior or concurrent 5-FU to the face allowed Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics Other: At least 30 days since prior megadoses of vitamins (e.g., more than 400 IU of vitamin E, 200 micrograms of selenium, or 1 g of vitamin C per day or more than the tolerable upper limits of any other supplement) At least 6 months since prior tretinoin to forearms Prior or concurrent tretinoin to the face allowed No concurrent mega-doses of vitamins No other concurrent investigational drug or device

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Alberts, MD, Study Chair — University of Arizona
Locations (1):
- Arizona Cancer Center, Tucson, Arizona, United States